CLINICAL TRIAL: NCT02099825
Title: Medication Enhanced Rapid Therapy
Acronym: MERiT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: COVID and staffing issues
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Eric Lenze, Professor of Psychiatry, Washington University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201306084
Record Dates: First submitted 2014-03-19; First posted 2014-03-31 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Anxiety Disorders
Keywords: adult male; anxiety; public speaking; healthy controls; exposure therapy; social anxiety; mifepristone; d-cycloserine
MeSH Terms: conditions — Anxiety Disorders; Speech | interventions — Cycloserine; Mifepristone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anxious Adult Males (Experimental): One time dosage of d-cycloserine and mifepristone at Session 2 prior to public speaking exposure sessions.
  Interventions: Drug: d-cycloserine and mifepristone
- Non-Anxious Adult Males (Active Comparator): One time dosage of d-cycloserine and mifepristone at Session 2 prior to public speaking exposure sessions.
  Interventions: Drug: d-cycloserine and mifepristone

INTERVENTIONS:
Drug: d-cycloserine and mifepristone — All participants will receive a one-time only dose of both, d-cycloserine and mifepristone at Session 2
  Other Names: mifepristone; Mifeprex; RU-486; one dose of up to 1200 mg; d-cycloserine; Seromycin; one dose of 250 mg

SUMMARY:
The purpose of this research study is to determine whether taking a one-time dose of a combination of putatively learning-enhancing medications can improve treatment response to a brief learning-based psychotherapy for public speaking anxiety. The two medications are (1) d-cycloserine (DCS), a medication that is an agonist (facilitator) of the NMDA glutamatergic receptor and has been shown in previous studies to facilitate some kinds of learning and memory; and (2) mifepristone, a medication that blocks cortisol, and in preclinical (animal) studies has been shown to reverse certain kinds of stress-related learning impairment or negative learning.

Specifically, the investigators goal is to determine if DCS and mifepristone taken together augment the learning that occurs during a brief psychotherapy session---a public speaking exposure exercise. Evidence for this learning effect would be a finding that participants have reduced anxiety at subsequent public speaking exposures.

DETAILED DESCRIPTION:
The study has a total of 4 visits, and the medications are given as a one-time dose at only one visit (the second visit).

1. During the first visit, a trained clinical interviewer will provide informed consent and conduct a structured clinical interview. Participants will be included if they are adult males diagnosed with social anxiety disorder and express a fear of public speaking, as well as approximately 10 healthy control participants. Eligible participants will be asked to complete self-report ratings of social anxiety and psychological symptoms and a standard interview about anxiety symptoms. The experimenter will conduct neuropsychological tests used to measure the participant's cognitive functioning.
2. At the second visit the participant will be administered a one-time only dosage of both medications. The participant will be asked to prepare a speech within a short period of time, this is an example of exposure therapy. In exposure therapy, people are exposed to a situation they fear, such as public speaking, in a safe and controlled environment. Often when people do exposure therapy, they find that the situations they have been afraid of are not actually as scary as they seem. The exposure exercise in this study will consist of giving a speech while being video-recorded. Before the exposure exercise, participants will be provided with 250mg DCS and up to 1200mg of mifepristone. Participants will rate their anxiety level and negative and positive affect before and after the speech, as well as during the speech. The experimenter will again conduct neuropsychological tests used to measure the participant's cognitive functioning.
3. (3) & (4) During the next two visits, participants will complete a second and third public speaking exposure exercise identical to the first, with the exception that they will NOT receive medication. Participants will complete a similar battery of symptom measures and anxiety ratings. The investigators will look at a change in anxiety ratings and symptomatology between exposure session 1, exposure session 2, and exposure session 3.

ELIGIBILITY:
For Potential Participants suffering from Social Anxiety Disorder or Social Phobia:

Inclusion Criteria:

* Male
* at least 18 years old
* current diagnosis of Social Anxiety Disorder or Social Phobia
* fear of public speaking
* medically stable and in good health
* if currently taking antidepressant treatment, must be on a stable dose for at least 8 weeks
* Liebowitz Social Anxiety Scale score of at least 30

Exclusion Criteria:

* Female
* inability to provide informed consent
* current or lifetime diagnosis of bipolar disorder, psychotic disorder or eating disorder
* current substance abuse or dependence within the last 6 months
* any cognitive, sensory, or communication problem that would prevent completion of the study
* severe mental health symptoms that require immediate treatment (i.e. active suicidality)
* current use of medication for diagnosis of one or more of the following: seizure disorder, kidney disease, liver disease
* current cancer (or history of metastatic cancer)
* current or recent use (within past 3 months) of systemic corticosteroids
* diabetic individuals
* untreated or unstable endocrinologic disease (i.e. hyperthyroidism)
* lifetime history of Cushing's disease or Addison's disease

For Control Group:

Inclusion Criteria:

* Male
* at least 18 years old
* no current diagnosis of Social Anxiety Disorder or Social Phobia
* reports no fear of public speaking
* Liebowitz Social Anxiety Scale score below or equal to 29

Exclusion Criteria:

* Female
* inability to provide informed consent
* current or lifetime diagnosis of bipolar disorder, psychotic disorder or eating disorder
* current substance abuse or dependence within the last 6 months
* any cognitive, sensory, or communication problem that would prevent completion of the study
* severe mental health symptoms that require immediate treatment (i.e. active suicidality)
* current use of medication for diagnosis of one or more of the following: seizure disorder, kidney disease, liver disease
* current cancer (or history of metastatic cancer)
* current or recent use (within past 3 months) of systemic corticosteroids
* diabetic individuals
* untreated or unstable endocrinologic disease (i.e. hyperthyroidism)
* lifetime history of Cushing's disease or Addison's disease

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-01-13 (Actual); Primary Completion 2022-10 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
Will measure medication tolerability and safety per participant report (i.e. few or no side effects severe enough to stop treatment) | End of Session 2--(7-10 days after Session 1)
  As measured by a self-reported side effects assessment conducted at this time point entitled: "Spontaneous Reports of Side Effects". This assessment will measure any reports of side effects as well as tolerability.

SECONDARY OUTCOMES:
Improvements in Anxiety as measured by several Self Report Assessments | Session 2- 1st exposure therapy session, occurs 7-10 days after Session 1
  Will measure CHANGES in anxiety level from 1st session to 2nd session as reported in the following self reports:
  Liebowitz Social Anxiety Scale (LSAS) Brief Resilient Coping Scale (BRCS) Post Event Processing Measure (PEP)-done at beginning of sessions 1, 3 and 4 (to reflect back on previous social engagements), and after speeches delivered at sessions 2, 3, and 4.
  Subjective Units of Distress Scale 0-100(SUDS 0-100) Social Interaction Anxiety Scale (SIAS) Social Phobia Scale (SPS) Subtle Avoidance Frequency Examination (SAFE) Positive and Negative Affect Scale (PANAS)
Level of Anxiety as measured by several Self Report Assessments | Session 1- initial self reports collected;
  Will measure initial anxiety level at Session 1 as reported in the following self reports:
  Liebowitz Social Anxiety Scale (LSAS) Brief Resilient Coping Scale (BRCS) Social Interaction Anxiety Scale (SIAS) Social Phobia Scale (SPS) Subtle Avoidance Frequency Examination (SAFE) Positive and Negative Affect Scale (PANAS)
Improvements in Anxiety as measured by several Self Report Assessments | Session 3- 2nd exposure therapy session- occurs 7- 10 days after Session 2
  Will measure CHANGES in anxiety level from 2nd session to 3rd session as reported in the following self reports:
  Liebowitz Social Anxiety Scale (LSAS) Brief Resilient Coping Scale (BRCS) Post Event Processing Measure (PEP)-done at beginning of sessions 1, 3 and 4 (to reflect back on previous social engagements), and after speeches delivered at sessions 2, 3, and 4.
  Social Interaction Anxiety Scale (SIAS) Social Phobia Scale (SPS) Subtle Avoidance Frequency Examination (SAFE) Positive and Negative Affect Scale (PANAS) Perception of Speech Performance (PSP)- done at beginning of sessions 3 and 4 (to reflect back on previous speech/ previous session), and after speeches delivered at sessions 2, 3, and 4.
  Subjective Units of Distress Scale 0-100(SUDS 0-100)
Improvements in Anxiety as measured by several Self Report Assessments | Session 4- 3rd exposure therapy- occurs 3 months later
  Will measure CHANGES in anxiety level from 3rd session to 4th session as reported in the following self reports:
  Liebowitz Social Anxiety Scale (LSAS) Brief Resilient Coping Scale (BRCS) Post Event Processing Measure (PEP)-done at beginning of sessions 1, 3 and 4 (to reflect back on previous social engagements), and after speeches delivered at sessions 2, 3, and 4.
  Social Interaction Anxiety Scale (SIAS) Social Phobia Scale (SPS) Subtle Avoidance Frequency Examination (SAFE) Positive and Negative Affect Scale (PANAS) Perception of Speech Performance (PSP)- done at beginning of sessions 3 and 4 (to reflect back on previous speech/ previous session), and after speeches delivered at sessions 2, 3, and 4.
  Subjective Units of Distress Scale 0-100(SUDS 0-100)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Lenze, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States